CLINICAL TRIAL: NCT05593484
Title: North STAR Trial: Specialty Telemedicine Access for Referrals (STAR) in Rural Alaska
Brief Title: School Screening and Telemedicine Specialty Referral to Address Childhood Hearing Loss in Rural Alaska
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Southcentral Foundation (Other); Duke University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 274168; R01DC020026 (NIH)
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Hearing Loss
Keywords: Rural; Hearing loss; Telemedicine; Telehealth; School; Disparities; Screening
MeSH Terms: conditions — Hearing Loss | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Approximately 23 schools from 3 regions are participating in the effectiveness trial. Clusters (~23 schools) will be randomized to one of two sequences. In academic year 2023-2024, all schools will receive enhanced screening (with standard referral). The Specialty Telemedicine Access for Referrals (STAR) intervention will be rolled out in a stepwise manner in academic years 2024-2025 and 2025-2026 depending on sequence randomization.
  Timeline update: Due to feedback from community partners, we extended the trial for one year. In academic year 2024-2025 all schools received the adapted enhanced screening. The STAR intervention will be rolled out in 2025-2026 and 2026-2027 depending on sequence randomization.
Who Masked: Outcomes Assessor
Masking Description: Statisticians will also be masked to group allocation until analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Referral (Other)
  Interventions: Other: Standard Referral
- Specialty Telemedicine Access for Referrals (STAR) (Other)
  Interventions: Other: Specialty Telemedicine Access for Referrals (STAR)

INTERVENTIONS:
Other: Standard Referral — Schools in the control condition will use standard referral, as determined by the school district. Standard referral is typically a letter home from the school to parents/caregivers of children who refer screening.
  Arms: Standard Referral
Other: Specialty Telemedicine Access for Referrals (STAR) — The STAR intervention will include a lay-friendly smartphone or tablet that connects to tools necessary for an ear and hearing evaluation. If a child requires referral from hearing screening, a school nurse/teacher will complete the established protocol for the STAR intervention and send the information asynchronously to an audiologist for review.
  Arms: Specialty Telemedicine Access for Referrals (STAR)

SUMMARY:
The prevalence of childhood hearing loss in rural Alaska is disproportionately high and predominately infection-related. With preventive screenings and access to health care, much of childhood hearing loss is preventable. Although state-mandated school screening helps identify children with hearing loss, loss to follow-up is pervasive and exacerbated by a scarcity of specialists in rural regions. A mixed methods cluster randomized trial conducted in northwest Alaska demonstrated that telemedicine can significantly reduce loss to follow-up. This stepped wedge trial, in partnership with Southcentral Foundation, will build on this existing work to develop a model that can be scaled in diverse environments.

We will adapt and implement a new telemedicine intervention called Specialty Telemedicine Access for Referrals (STAR). This trial will be conducted in 3 regions in rural Alaska that represent multiple healthcare systems. Based on stakeholder feedback and evidence generated from the previous trial, an enhanced mobile health (mHealth) hearing screening will be implemented in all participating schools prior to the STAR intervention, and the telemedicine referral to specialty care (STAR intervention) will be moved from the clinic directly into the school.

This stepped-wedge cluster randomized trial is part of a larger hybrid type 1 effectiveness-implementation trial. The stepped wedge trial will evaluate the effectiveness of the STAR intervention in reducing loss to follow-up from referred school hearing screening in 3 regions of Alaska: Kodiak, Petersburg and Lower Yukon (n=23 schools, ~2,015 K-12 students/year). The STAR Intervention will be compared to the standard referral of a letter home to families. Cluster randomization at the level of school will be performed, with schools (clusters) randomized to one of two sequences. The effectiveness outcome (i.e., proportion of children who receive follow-up) will be evaluated over three academic years (2023-2026), with STAR rolled out in a stepwise manner for each of the two sequences (academic year 2024-2025 for sequence 1 and academic year 2025-2026 for sequence 2). The control periods for each sequence will be academic year 2023-2024 for sequence 1 and academic years 2023-2024 and 2024-2025 for sequence 2. Enhanced screening will be rolled out to both sequences at the same time (i.e., non-randomized) beginning academic year 2023-2024. An implementation evaluation will be conducted to refine and adapt the enhanced hearing screening and STAR intervention throughout the trial. Implementation data will be collected starting academic year 2022-2023 and then annually for each of the subsequent years.

Timeline update: Based on feedback from community partners, we extended the trial for one year to allow for community-informed adaptations of the enhanced screening. Now the STAR intervention will be rolled out in 2025-2026 for sequence 1 and 2026-2027 for sequence 2.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in one of the participating schools in the 3 regions
* Children from grades (K-12) that are typically screened within participating schools
* Eligible regardless of age, gender, race, or ethnicity

Exclusion Criteria:

N/A

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8060 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of children who receive follow-up | Proportion of children who receive follow-up will be measured by the occurrence of an ear/hearing encounter, up to 60 days from the date of screening.
  This outcome will be measured each school year, for 4 years, based on the updated timeline.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hirschfeld, MD,PhD, Principal Investigator — Vice President-Specialty Services, Southcentral Foundation, Alaska Native Medical Center; Susan Emmett, MD, MPH, Principal Investigator — University of Arkansas Medical Sciences
Locations (1):
- Southcentral Foundation, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Yes
This study focusses on population outcomes. School and health data will remain with local education and healthcare entities, and the study team will receive deidentified information. Data sharing will be considered upon request pending appropriate local approval.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Robler SK, Bettger JP, Turner E, Platt A, Arthur D, Hofstetter P, Lane H, Srinivasan T, Deshpande S, Hirschfeld M, Emmett SD. School-based enhanced hearing screening and specialty telehealth follow-up for hearing loss among children in rural Alaska: study protocol for a hybrid effectiveness-implementation stepped wedge, cluster-randomized controlled trial (North STAR trial). Trials. 2025 May 27;26(1):175. doi: 10.1186/s13063-025-08864-0. PMID 40426213
- [Derived] Robler SK, Bettger JP, Turner E, Platt A, Arthur D, Hofstetter P, Lane H, Srinivasan T, Deshpande S, Hirschfeld M, Emmett SD. School-Based Enhanced Hearing Screening and Specialty Telehealth Follow-Up for Hearing Loss Among Children in Rural Alaska: Study Protocol for a Hybrid Effectiveness-Implementation Stepped Wedge, Cluster-Randomized Controlled Trial (North STAR Trial). Res Sq [Preprint]. 2025 Apr 1:rs.3.rs-5252346. doi: 10.21203/rs.3.rs-5252346/v1. PMID 40235498